CLINICAL TRIAL: NCT06690892
Title: Understanding the Cognitive and Brain Health Effects of Increasing Beef Consumption in Young Adults
Brief Title: Investigating the Effects of Beef Consumption on Cognitive and Brain Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23404
Record Dates: First submitted 2024-10-28; First posted 2024-11-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dietary Intervention; Dietary Proteins; Dietary Assessment; Cognitive Ability, General
Keywords: beef consumption; beef dietary intervention; brain health; cognitive health
MeSH Terms: interventions — Freezing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will participate in the 12-week beef dietary intervention study. Participants will be provided with 5 portions of ready-to-eat beef in frozen packages per week, and consume 5 portions per week. Each portion of beef provided to this group will weigh 5 ounces.
  Interventions: Dietary Supplement: Ready-to-eat beef in frozen, 5-oz packages
- Control Group (Placebo Comparator): The control group will participate in the 12-week beef dietary intervention. Participants will be provided with 5 portions of ready-to-eat beef in frozen packages per week, and consume 5 portions per week. Each portion of beef provided to this group will weigh 1 ounce.
  Interventions: Dietary Supplement: Ready-to-eat beef in frozen, 1-oz packages

INTERVENTIONS:
Dietary Supplement: Ready-to-eat beef in frozen, 5-oz packages — The dietary intervention lasts 12 weeks for each individual. Participants in the experimental group will receive this intervention. Each participant will acquire 5 portions of ready-to eat beef in frozen packages per week, and consume 5 portions per week (1 portion of sirloin cap steak strips, 1 portion of shredded chuck roast, 1 portion of petite shoulder medallions, and 2 portions of ground beef crumbles); each portion of ready-to-eat beef in this intervention will weigh 5 ounces.
  Arms: Experimental Group
Dietary Supplement: Ready-to-eat beef in frozen, 1-oz packages — The dietary intervention lasts 12 weeks for each individual. Participants in the control group will receive this intervention. Each participant will acquire 5 portions of ready-to eat beef in frozen packages per week, and consume 5 portions per week (1 portion of sirloin cap steak strips, 1 portion of shredded chuck roast, 1 portion of petite shoulder medallions, and 2 portions of ground beef crumbles); each portion of ready-to-eat beef in this intervention will weigh 1 ounce.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if eating more beef will lead to better cognition and a healthier brain in younger adults. The main questions it aims to answer are:

* Does eating more beef lead to higher scores on cognitive tests and better quality of life?
* Does eating more beef lead to better brain function?

Researchers will compare participants in the experimental group (participants who will eat 25 ounces of beef every week during the dietary intervention) to control participants (participants who will eat 5 ounces of beef every week during the dietary intervention).

Participants will:

* Be instructed to prepare and consume ready-to-eat beef meals along with their regular diet and not eat any more beef other than what they are given
* Visit the study facilities once every week to pick up ready-to-eat beef meals; and complete a brief survey every week to track their consumption of the provided beef meals, and a dietary survey every 4 weeks
* Visit the study facilities before and after the 12-week of intervention period for researchers to study them

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effects of beef consumption on cognitive and brain health in healthy younger adults. Specifically, we seek to evaluate the effects of beef consumption on measures of executive function, memory, psychological well-being, and sleep quality. Additionally, we will explore the effects of increased beef consumption on measures of brain health derived from structural and functional brain imaging.

The study will consist of two groups of participants: experimental and control. Participants from both groups will take part in a 12-week dietary intervention. Throughout the intervention, participants in the experimental group will receive 5 portions of ready-to-eat lean beef in frozen packages every week; and consume 5 portions per week. Each serving of ready-to-eat beef for the experimental group will weigh 5-ounces. Participants in the control group will also receive 5 portions of ready-to-eat lean beef in frozen packages every week; and consume 5 portions per week. Each serving of ready-to-eat beef for the control group will weigh 1-ounce. Study compliance will be evaluated through weekly surveys about beef consumption.

In addition, all participants will complete pre- and post-intervention assessments:

* MRI scan, including structural and functional brain imaging
* a comprehensive questionnaire battery evaluating cognitive and psychological measures
* neuropsychological tasks
* a blood draw

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Males and females; Age 19-24
* Willingness to adhere to the ready-to-eat beef intervention regimen
* Enrolled at University of Nebraska-Lincoln
* BMI between 18.5 and 39.9
* Not pregnant or nursing
* No history of cognitive or metabolic diseases indicated by diagnosis, including neurodegenerative disease, stroke, Type 1 and 2 diabetes, metabolic syndrome, cardiovascular disease, liver disease, kidney disease, and cancer
* No history of eating or anxiety disorders
* Willing to discontinue dietary supplement use throughout the duration of the study, if they are consuming supplement at the time of the registration
* No known contraindication to MRI scans as determined by the MRI screening survey questions

Exclusion Criteria:

* Current use of medications that may affect their responses to dietary intervention, such as amphetamines, antidepressants, anti-diabetic medications, laxatives, antibiotics, statins and diuretics.
* Known intolerance or allergy to beef
* Current use of nicotine products, including vaping
* Previous use of nicotine products, including vaping, within the recent 6 months at the time of pre-screening

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
WAIS-V | Baseline and after 12 weeks
  Wechsler Adult Intelligence Scale, verison 5. Comprehensive assessment battery for measuring cognitive abilities
NIH Toolbox (Dimensional Change Card Sort) | Baseline and after 12 weeks
  Test for executive function and cognitive flexibility
NIH Toolbox (Flanker) | Baseline and after 12 weeks
  test for executive functions: attention and inhibitory control
NIH Toolbox (List Sorting Working Memory Test) | Baseline and after 12 weeks
  Test for working memory
Cognitive Reflection Test | Baseline and after 12 weeks
  Test to measure the ability to suppress an intuitive wrong answer in favor of a more reflective correct answer
Short Form-36 Health Survey | Baseline and after 12 weeks
  self-report measure of health status and quality of life
Decision Outcome Inventory | Baseline and after 12 weeks
  an assessment of outcomes of real-life decisions
Pittsburgh Sleep Quality Index | Baseline and after 12 weeks
  Self-report assessment of sleep quality over the past month. The survey includes measures related to Sleep Latency, Sleep Duration, Sleep Efficiency, Sleep Disturbances, Use of Sleep Medications, Daytime Fatigue, and Sleep Quality
Symptom Checklist 90-Revised | Baseline and after 12 weeks
  self-report assessment of psychological symptoms related to the domains of somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism

SECONDARY OUTCOMES:
Brain Imaging | Baseline and after 12 weeks
  * T1- weighted imaging to visualize the structure of the brain
  * Functional MRI of the whole brain to examine changes in brain activity and functional topology
  * Diffusion tensor imaging to map the white matter structures in the brain

OTHER OUTCOMES:
Height | Baseline and after 12 weeks
  measured in feet and inches
Weight | Baseline and after 12 weeks
  measured in pounds (lbs)
Body Mass Index | Baseline and after 12 weeks
  Calculated by body mass divided by the square of the body height, unit in kg/m^2
Heart Rate | Baseline and after 12 weeks
  Heart rate will be reported as beats per minute.
Systolic and Diastolic Blood Pressure | Baseline and after 12 weeks
  Measured in mmHg
Body Composition | Baseline and after 12 weeks
  Body composition will be measured in body fat%
Grip Strength | Baseline and after 12 weeks
  Participants will squeeze a hydraulic device three times with their right hand. Grip strength will be obtained by averaging the three measurements, which will be measured in kilograms.
Blood-based biomarkers associated with consumption of beef | Baseline and after 12 weeks
  Biomarkers under evaluation include inflammatory biomarkers and nutrient biomarkers in blood from participants

CONTACTS AND LOCATIONS:
Overall Officials: Aron Barbey, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Study findings will be submitted to peer-reviewed journals such as those that follow the ICMJE's recommendations for the Conduct, Reporting, Editing and Publication of Scholarly Work in Medical Journals. The data collected in this project may be shared through public-use files, repositories or other means outside of the approved research team as a requirement of publication. All data will be identified with subject IDs only when shared. Research records such as informed consent forms, MRI Safety Screening forms, research compliance records, masterlist linking names to subject IDs will not be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: IPD and supporting information will be available beginning 1 year after the publication of results with no end date.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access the IPD and supporting information. Researchers are not restricted on the type of analyses, as long as they are methodologically sound. The statistical methods for those analyses must be approved before the researchers can gain access to the data.
  For data sharing, a proposal that describes planned analyses must be submitted to the study's contact personnel for review. A data sharing agreement must be signed between the institution of the requesting researchers and the institution of the study's principal investigator.

REFERENCES:
- [Background] Zhang H, Hardie L, Bawajeeh AO, Cade J. Meat Consumption, Cognitive Function and Disorders: A Systematic Review with Narrative Synthesis and Meta-Analysis. Nutrients. 2020 May 24;12(5):1528. doi: 10.3390/nu12051528. PMID 32456281
- [Background] Hepsomali P, Groeger JA. Diet and general cognitive ability in the UK Biobank dataset. Sci Rep. 2021 Jun 3;11(1):11786. doi: 10.1038/s41598-021-91259-3. PMID 34083695